CLINICAL TRIAL: NCT05389475
Title: Anoplasty for Post Hemorroidectomy Anal Stenosis : Diamond Versus V-Y Flap Techniques
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Mokbel, doctor, Assiut University
Other Study IDs: Diamond flap
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Anoplasty in Treatment of Post Hemorroidectomy Anal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: anoplasty in treatment of post hemorroidectomy anal stenosis — Diamond flap versus V-Y flap

SUMMARY:
The aim of the study to evaluate the outcome of diamond flap versus V-Y flap for treatment of severe post hemorroidectomy anal stenosis .

DETAILED DESCRIPTION:
Anal stenosis is diagnosed when there is a narrowing of the anal canal and subsequent loss of normal elasticity that makes its wall rigid and unable to be dilated to permit normal pain-free defecation(1). The underlying pathology of anal stenosis results from a wide variety of either functional or anatomical causes . In functional anal stenosis, the presence of a hypertonic internal anal sphincter is the major cause of the narrowing, whereas in anatomical anal stenosis, the normal elastic anoderm replaced by an inelastic rigid fibrous tissue is the major cause of the anal canal narrowing(2). The best way of treatment of anal stenosis is avoiding its occurrence, as the major cause is following surgical hemorrhoidectomy, particularly when a large area of anoderm lining the anal canal is removed during the operation, but can also complicates other anorectal surgical operations(3). The patient usually experiences painful defecation, incomplete evacuation, pellet stool, or rectal bleeding. These manifestations force the patient to rely on daily laxatives or enemas in bowel evacuation(1). Usually physical examination is all that is needed to confirm the diagnosis of anal stenosis, including inspection of the anal canal, perianal skin, and digital rectal examination]. Anatomical anal stenosis can be classified according to Milsom and Mazie (4) based on the severity of the anal canal narrowing into mild anal stenosis, when the anal canal can be examined by a well-lubricated index finger or a medium-sized Hill-Ferguson retractor; moderate anal stenosis, when forceful dilatation is required to insert either the index finger or a medium-sized Hill-Ferguson retractor; and severe anal stenosis, when neither the little finger nor a small-sized Hill-Ferguson retractor can be inserted.

In most patients with mild to moderate anal stenosis, medical management with stool softeners or fiber supplements , emollient laxatives , high fiber diet to help softener of stool and make it pass easily would be a choice(5).

However, different surgical procedures are reserved for patients with severe anal stenosis and in case of failed medical treatment. The choice of the most appropriate procedure is based on the severity where lateral sphincterotomy could be sufficient for a patient with a mild and sometimes moderate degree of anal stenosis after failure of medical treatment(6). However, various flap anoplasty procedures should be reserved for the more severe cases to replace the cicatrized tissues The aim of various techniques of anoplasty is to restore the normal function of the narrowed anal canal by dividing the stricture, and this leads to widening of the anal canal while preserving the anal continence and thus pain-free bowel evacuation(7).

Prevention The best treatment for anal stenosis after hemorrhoidectomy is a meticulous approach in the operating room during the primary operation. The risk of anal stenosis increases with the complexity and extent of the hemorrhoids treated. Surgical therapy of extensive and complicated hemorrhoids should only be approached by surgeons experienced in this operation. The keys to prevention of anal stenosis after hemorrhoidectomy are meticulous submucosal dissection with avoidance of injury to the internal sphincter muscle and the preservation of sufficient intact anoderm between excision sites, generally considered at least 1 cm of intact intervening anoderm. Additionally, limiting the number of hemorrhoids excised in a given setting will also help to limit the incidence of postoperative stenosis. Nonoperative Intervention The cornerstone of therapy for anal stenosis from all causes is dietary modification, including a combination approach utilizing stool softeners as well as increased fiber intake and water consumption. For many patients with mild stenosis, these simple measures may alleviate the patient's symptoms. For patients not initially responsive to these measures, and those with moderate steno ses, it is reasonable to attempt a course of manual dilation in addition to the above measures. This program consists of an initial dilation in the operating room or clinic, if tolerated, followed by serial dilations at home by the patient using either a finger or a dilator. This can be facilitated and better tolerated through the use of anesthetic jelly (e.g., lidocaine 2%). The majority of patients with mild stenosis will achieve symptom alleviation with this approach, as will many patients with moderate stenosis. Manual dilation does have some risks, such as perforation, but these risks are low

Surgical methods in treatment of anal stenosis contain:

1. Lateral Internal Sphincterotomy
2. Lateral Mucosal Advancement Flap
3. V-Y Advancement Flap
4. Diamond-Shaped Flap
5. House Flap
6. U-shaped Flap

ELIGIBILITY:
Inclusion Criteria:

* Patients with post-surgical severe anal stenosis based on Milsom and Mazier classification after the failure of non-operative measures were included.

Exclusion Criteria:

* (1) Patients with functional stenosis as acute anal fissure. (2) Patients with a recent history of anal stenosis who had no medical treatment trial.

  (3) Patients with mild or moderate anal stenosis who expected to respond to medical treatment.

  (4) Patients with inflammatory bowel disease, tuberculosis, or perianal fistula.

  (5) Patients with previous radiotherapy or previous anal malignancy. (6) Patients with previous anoplasty.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Based on determining the main outcome variable, the estimated minimum required sample size is 52cases (26in each group).
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
comparison between outcomes of Diamond flap versus V-Y flap in treatment of anal stenosis post hemorroidectomy | 3 months
  Postoperative complication as anal pain , bleeding , infection , healing , incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Momen Shalqamy, PhD, Study Director — Moamen.shalkamy@aun.edu.eg; Gamal Abdelhamid, PhD, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] 1 Liberman H, Thorson AG. How I do it: anal stenosis. Am J Surg 2000; 179:325-329. 2 Casadesus D, Villasana LE, Diaz H, Chavez M, Sanchez IM, Martinez PP, et al. Treatment of anal stenosis: a 5-year review. ANZ J Surg 2007:557-559. 3 Caplin DA, Kodner IJ. Repair of anal stricture and mucosal ectropion by simple flap procedures. Dis Colon Rectum 1986; 29:92-94. 4 Milsom JW, Mazier WP. Classification and management of postsurgical anal stenosis. Surg Gynecol Obstet 1986; 163:60-64. 5 Corman ML, Bergamaschi RCM, Nicholls RJ, Turnbull FRBJr, editors. Corman's colon and rectal surgery. 6th ed. New York: Stony Brook University 2013. 327. 6 Owen HA, Edwards DP, Khosraviani K, Phillips RK. The house advancement anoplasty for treatment of anal disorders. J R Army Med Corps 2006; 152:87-88. 7 Duieb Z, Appu S, Hung K, Nguyen H. Anal stenosis: use of an algorithm to provide a tension-free anoplasty. ANZ J Surg 2010; 80:337-340. 778 The Egyptian Journal of Surgery, Vol. 39 No. 3, July-September 2020 [Downloaded free from http://www.ejs.eg.net on Sunday, October 10, 2021, IP: 197.36.13.202] 8 Maria G, Brisinda G, Civello IM. Anoplasty for the treatment of anal stenosis. Am J Surg 1998; 175:158-160 9 Brisinda G. How to treat hemorrhoids. Prevention is best; hemorrhoidectomy needs skilled operators. BMJ 2000; 321:582-583. 10 Shevchuk IM, Sadoviy IY, Novytskiy OV. Surgical treatment of postoperative stricture of anal channel. Klin Khir 2015; 9:20-22. 11 Giordano P, Gravante G, Grondona P, Ruggiero B, Porrett T, Lunniss PJ. Simple cutaneous advancement flap anoplasty for resistant chronic anal fissure: a prospective study. World J Surg 2009; 33:1058-1063. 12 Abr-Gama A, Sobrado CW, Araujo SE, Nahas SC, Birbojm I, Nahas CS, et al. Surgical treatment of anal stenosis: assessment of 77 anoplasties. Clinics 2005; 60:17-20. 13 Nelson R. Operative procedure for fissure in ano. Cochrane Database Syst Rev 2005; 9:C D002199. 14 Carditello A, Milone A, Stilo F, Mollo F, Basile M. Surgical treatment of anal stenosis following hemorrhoid surgery. Results of 150 combined mucosal advancement and internal sphincterotomy. Chir Ital 2002; 54:841-844. 15 Brisinda G, Vanella S, Cadeddu F, Marniga G, Mazzeo P, Brandara F, Maria G. Surgical treatment of anal stenosis. World J Gastroenterol 2009; 15:1921-1928. 16 Aitola PT, Hiltunen KM, Matikainen MJ. Y-V anoplasty combined with internal sphincterotomy for stenosis of the anal canal. Eur J Surg 1997; 163:839-842